CLINICAL TRIAL: NCT03525418
Title: Lomecel-B Injection in Patients With Hypoplastic Left Heart Syndrome: A Phase I/II Study (ELPIS)
Brief Title: Lomecel-B Delivered During Stage II Surgery for Hypoplastic Left Heart Syndrome (ELPIS)
Acronym: ELPIS
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Longeveron Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00-0000-05
Record Dates: First submitted 2018-02-19; First posted 2018-05-15 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: HLHS
Keywords: Pediatrics

STUDY DESIGN:
Intervention Model Description: Phase 1: 10 patient safety run-in: all patients treated with LMSCs during Stage II surgery.
  Phase 2: 20 patients randomized 1:1 to receive either LMSCs or no cells (controls) during Stage II surgery.
Who Masked: Participant, Investigator
Masking Description: Phase 1: no masking. Phase 2: HLHS patients which will be randomized to the treatment and control arms in a 1:1 ratio
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A - Phase 1 (Open Label) (Experimental): 10 consecutive HLHS patients will be enrolled and treated with Longeveron Mesenchymal Stem Cells (LMSCs). A single administration of LMSCs will be performed via intramyocardial injections during the Stage II (BDCPA) surgery. Dosing is based on body weight. Each LMSC-treated patient will be given 2.5 x 105 LMSCs per kg of body weight. The entire dose of the cells will be roughly 600 microliters.
  Interventions: Biological: Longeveron Mesenchymal Stem Cells
- Cohort B - Phase 2 Treatment Group (Experimental): Double-blinded, in which 20 HLHS patients will be randomized to either receive treatment with Longeveron Mesenchymal Stem Cells (LMSCs) (Cohort B, 10 patients) performed via intramyocardial injections during the Stage II (BDCPA) surgery, or will receive no cells and no injection (Cohort C, 10 patients) during the Stage II (BDCPA) surgery. The second stage is to obtain preliminary safety and efficacy data the will enable and guide a subsequent larger Phase 2 trial.
  Interventions: Biological: Longeveron Mesenchymal Stem Cells
- Cohort C - Phase 2 Control Group (No Intervention): Double-blinded, in which 20 HLHS patients will be randomized to either receive treatment with Longeveron Mesenchymal Stem Cells (LMSCs) (Cohort B, 10 patients) performed via intramyocardial injections during the Stage II (BDCPA) surgery, or will receive no cells and no injection (Cohort C, 10 patients) during the Stage II (BDCPA) surgery. The second stage is to obtain preliminary safety and efficacy data the will enable and guide a subsequent larger Phase 2 trial.

INTERVENTIONS:
Biological: Longeveron Mesenchymal Stem Cells — Allogeneic bone marrow-derived mesenchymal stem cell
  Other Names: LMSCs
  Arms: Cohort A - Phase 1 (Open Label); Cohort B - Phase 2 Treatment Group

SUMMARY:
This study is designed to assess the safety, tolerability, and efficacy of Lomecel-B as an adjunct therapy to the standard stage II (BDCPA) surgical intervention for HLHS. Lomecel-B will be delivered via intramyocardial injections

DETAILED DESCRIPTION:
This study is designed to assess the safety, tolerability, and efficacy of Lomecel-B (formerly LMSCs) as an adjunct therapy to the standard stage II (BDCPA) surgical intervention for HLHS, which is typically performed at 4 - 6 months after birth. Lomecel-B will be delivered via intramyocardial injections.

A total of 30 patients will be enrolled in 2 stages with 3 Cohorts.

In the first stage, 10 consecutive HLHS patients will be enrolled and treated with Lomecel-B (Cohort A). The first 3 patients will be treated no less than 5 days apart, and will be evaluated for any treatment-emergent adverse events (TE-AEs) (e.g., induced myocardial infarction or perforation). These patients will undergo full evaluation for 5 days to demonstrate safety prior to proceeding with the remainder of the cohort. After 6 months post-treatment of the last patient of Cohort A, a formal safety review will be conducted prior to proceeding to the next phase.

The second stage is double-blinded, in which 20 HLHS patients will be randomized to either receive treatment with Lomecel-B (Cohort B, 10 patients), or will receive no cells and no injection (Cohort C, 10 patients).

ELIGIBILITY:
Inclusion Criteria: all patients must have HLHS (all types) requiring BDCPA surgery.

Exclusion Criteria: all patients must not have any of the following.

1. Significant coronary artery sinusoids.
2. Requirement for mechanical circulatory support prior to BDCPA surgery.
3. Underlying evidence of arrhythmia requiring anti-arrhythmia therapy.
4. Need for concomitant surgery for aortic coarctation or tricuspid valve repair.
5. HLHS and restrictive or intact atrial septum.
6. Undergoing the Stage I (Norwood) procedure that does not have HLHS.
7. Serum positivity for: HIV; hepatitis B virus surface antigen (HBV BsAg); and/or viremic hepatitis C virus (HCV).
8. Parent/guardian that is unwilling or unable to comply with necessary follow-up.
9. Unsuitability for the study based on the Investigator's clinical opinion.
10. Documented chromosomal abnormalities

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety: To evaluate the safety and feasibility of intramyocardial injection of LMSCs during the Stage II (BDCPA) operation for HLHS via incidence of Treatment-Emergent Serious Adverse Events. | Evaluated through 1 year post-treatment.
  The incidence of Treatment-Emergent Serious Adverse Events will be evaluated, including: sustained/symptomatic ventricular tachycardia requiring intervention with inotropic support; aggravation of heart failure; myocardial infarction; unplanned cardiovascular operation for cardiac tamponade; infection during the first month post-treatment; and death.

SECONDARY OUTCOMES:
Efficacy: Change from baseline in right ventricular ejection fraction (%). | Evaluated through 1 year post-treatment.
  Used to assess cardiac function.
Efficacy: Change from baseline in right ventricular end-systolic volume. | Evaluated through 1 year post-treatment.
  Used to assess cardiac function.
Efficacy: Change from baseline in right ventricular end-diastolic volume. | Evaluated through 1 year post-treatment.
  Used to assess cardiac function.
Efficacy: Change from baseline in right ventricular end-diastolic diameter. | Evaluated through 1 year post-treatment.
  Used to assess cardiac function.
Efficacy: Change from baseline tricuspid regurgitation. | Evaluated through 1 year post-treatment.
  Used to assess cardiac function. Measured by serial echocardiograms and MRI.
Efficacy: Change in weight (in kilograms). | Evaluated through 1 year post-treatment.
  Used to assess change in somatic growth.
Efficacy: Change in height (in centimeters). | Evaluated through 1 year post-treatment.
  Used to assess change in somatic growth.
Efficacy: Change in head circumference (in centimeters). | Evaluated through 1 year post-treatment.
  Used to assess change in somatic growth.
Efficacy: Number of patients with Treatment-Emergent Adverse Events, and total number of occurrences of Treatment-Emergent Adverse Events, through-out participation in trial. | Evaluated through 1 year post-treatment.
  Treatment-Emergent Adverse Events will be assessed via incidence of co-morbidity, which include: cardiovascular morbidity; need for transplantation; re-hospitalizations; cardiovascular mortality; and all-cause mortality.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Emory University/Childen's Healthcare of Atlanta, Atlanta, Georgia
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins University Hospital, Baltimore, Maryland
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Utah/Heart Center-Primary Children's Hospital, Salt Lake City, Utah

REFERENCES:
- [Derived] Kaushal S, Hare JM, Hoffman JR, Boyd RM, Ramdas KN, Pietris N, Kutty S, Tweddell JS, Husain SA, Menon SC, Lambert LM, Danford DA, Kligerman SJ, Hibino N, Korutla L, Vallabhajosyula P, Campbell MJ, Khan A, Naioti E, Yousefi K, Mehranfard D, McClain-Moss L, Oliva AA, Davis ME. Intramyocardial cell-based therapy with Lomecel-B during bidirectional cavopulmonary anastomosis for hypoplastic left heart syndrome: the ELPIS phase I trial. Eur Heart J Open. 2023 Jan 11;3(2):oead002. doi: 10.1093/ehjopen/oead002. eCollection 2023 Mar. PMID 36950450